CLINICAL TRIAL: NCT03721562
Title: Antibiotic Resistance in Global Pediatric Oncology Centers
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Johns Hopkins University (Other); Tarleton State University (Unknown)
Responsible Party: Sponsor
Other Study IDs: ARGO
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Antibiotic Resistant Infection
Keywords: Antibiotic Resistance; Gram Negative Bacteria; Pediatric Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antibiotic resistance is one of the major health threats facing global as well as domestic populations, however it is not well characterized in pediatric patients. Pediatric patients receiving cancer-directed therapy have several risk factors implicated in development of antibiotic resistance including multiple courses of antibiotics, repeated exposures to the hospital environment, indwelling devices and chemotherapy-related damage to mucosal barriers. The investigators propose to capitalize upon the unique position of St. Jude Global within the global pediatric oncology community by using its regional alliance network to describe the molecular epidemiology of antibiotic resistance in Gram-negative bacteria in this population.

Primary Objectives

1. Describe the epidemiology and the phenotypic and previously determined molecular determinants of antimicrobial resistance in Gram-negative organisms isolated from pediatric diagnostic specimens in selected Central American and US sites with capacity to treat pediatric cancer
2. Utilize strain typing by whole genome sequencing to describe relatedness between organisms at participating sites

DETAILED DESCRIPTION:
Participating clinical microbiology laboratories will flag any Gram-negative bacteria meeting inclusion criteria. Bacteria will be subcultured; one sample will be lysed and shipped to St. Jude; the remaining sample will be stored onsite for the duration of the study. Samples of bacteria from both oncology and non-oncology patients will be included. Whole genome sequencing will be performed on the bacterial samples at St. Jude and the genotypic and phenotypic antimicrobial resistance testing (AST) results compared. Genotypic results will additionally be used to describe phylogenetic relationships and potential transmission events both within and between sites.

Each participating location will collect limited clinical data corresponding to disease and treatment related factors on the affected patient. This will include sociodemographic variables, oncologic diagnosis, treatment phase, presence of a central venous catheter or other foreign body, antibiotic treatment within the past month, and previous history of colonization or infection by a resistant organism.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric (0-18 years of age) patients having a bacteria isolated from a sterile site (blood, cerebrospinal fluid, body fluid) or urine positive for a Gram-negative bacteria nonsusceptible to at least 1 of the following: third generation cephalosporin, fourth generation cephalosporin or carbapenem OR screening positive for carbapenemase or extended spectrum beta lactamase (ESBL) production.

Exclusion Criteria:

* Repeated isolation of the same organism from the same patient within the study period.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric (0-18 years of age) patients having a bacteria isolated from a sterile site (blood, cerebrospinal fluid, body fluid) or urine positive for a Gram-negative bacteria nonsusceptible to at least 1 of the following: third generation cephalosporin, fourth generation cephalosporin or carbapenem OR screening positive for carbapenemase or extended spectrum beta lactamase (ESBL) production.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Patterns of organism and resistance in participating sites | approximately 6 months after completion of data collection
  Number of isolated organisms by anatomic site and geographic site
Patterns of organism and resistance in participating sites | approximately 6 months after completion of data collection
  Number of antibiotic resistance genes/mutations of interest by geographic site
Patterns of organism and resistance in participating sites | approximately 6 months after completion of data collection
  Correlation of known mutations/genes of interest with drug resistance phenotype
Genetic relatedness between bacteria at participating sites | approximately 6 months after completion of data collection
  Whole genome sequencing results will be used to describe whether isolated organisms appear to be related phylogenetically.

CONTACTS AND LOCATIONS:
Overall Officials: Sheena Mukkada, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (5):
- United States (2):
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
- Hospital Nacional de Niños Benjamín Bloom, San Salvador, El Salvador
- Unidad Nacional de Oncología Pediátrica, Guatemala City, Guatemala
- Hospital del Niño, Panama City, Panama

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols